CLINICAL TRIAL: NCT00409110
Title: Relationship Between Ocular Pulse Amplitude And Choroidal Laser Doppler Flowmetry In Healthy Subjects
Brief Title: Ocular Pulse Amplitude And Choroidal Laser Doppler Flowmetry
Status: Terminated | Type: Observational
Why Stopped: methodological problems
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orguel, University Hospital, Basel, Switzerland
Other Study IDs: 082-KAR-2006-001
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: Ocular Pulse Amplitude; Dynamic Contour Tonometry; Pulsatility Index; Choroidal Laser Doppler Flowmetry; Finometer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study intends to investigate the relationship between choroidal blood flow and ocular pulse amplitude (OPA).

DETAILED DESCRIPTION:
One eye is randomly selected in 18 healthy subjects. OPA is assessed with Dynamic Contour Tonometry. Submacular choroidal blood flow is measured with Laser Doppler Flowmetry. During both examinations the systemic blood pressure is continuously recorded with Finometer. An average systolic and diastolic LDF parameter flow during 30 seconds are determined and the pulsatility index is calculated according to the formula (LDFsys-LDFdia)/LDFdia. An association of OPA with the LDF pulsatility index, systemic blood pressure values and mean intraocular pressure will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects should present no history of ocular diseases, of current topical medication, or of drug or alcohol abuse. Furthermore, a best corrected visual acuity above 20/25 in both eyes, lack of pathological findings upon a slit-lamp examination and dilated direct fundoscopy, and an IOP < 21 mmHg in both eyes will be required.

Exclusion Criteria:

* History of chronic or recurrent severe inflammatory eye disease such as scleritis or uveitis.
* History of ocular trauma or intraocular surgery. History of infection or inflammation within the past 3 months.
* History and clinical evidence for other retinal disease such as age-related degeneration, or diabetic retinopathy.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
An association of OPA with the LDF pulsatility index | 30 seconds

SECONDARY OUTCOMES:
An association of OPA with the systemic blood pressure values | 30 seconds
An association of OPA with mean intraocular pressure | 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orguel, MD, Study Director — University Eye Clinic Basel
Locations (1):
- University Eye Clinic Basel, Basel, Canton of Basel-City, Switzerland